CLINICAL TRIAL: NCT00734383
Title: PRO-TECT II: Propofol Cardioprotection for Type II Diabetics
Brief Title: Propofol Cardioprotection for Type II Diabetics
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H04-70456
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Myocardial Injury
Keywords: coronary artery bypass surgery; coronary artery bypass grafting; cardiopulmonary bypass; diabetes; myocardial injury markers,; sex differences; cardiac anesthesia; inhalational anesthetics
MeSH Terms: conditions — Diabetes Mellitus | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Propofol Cardioprotection
  Interventions: Drug: Propofol
- 2 (Experimental): Volatile Anesthesia Preconditioning
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Propofol cardioprotection : Ten minutes prior to initiation of CPB, we will stop delivery of isoflurane, inject 1 mg/kg iv and then continuously infuse propofol at 120µg/kg/min IV until 15 min after release of the aortic cross clamp (reperfusion).
  Arms: 1
Drug: Propofol — Volatile Anesthetic preconditioning : Anesthesia will be maintained using an inspired concentration of isoflurane between 0.5-2% before, during, and after CPB, without administration of propofol. For ten minutes prior to the initiation of CPB we will deliver Isoflurane 2.5% end tidal then resume maintenance anesthesia as described.
  Arms: 2

SUMMARY:
The purpose of this study is to determine if an intravenous anesthetic with antioxidant properties will protect the heart of diabetic patients from injury while undergoing coronary bypass surgery.

DETAILED DESCRIPTION:
Diabetic patients are at elevated risk for low cardiac output syndrome. This high risk scenario adversely affects up to 26% of patients recovering from cardiac surgery. Aggressive hemodynamic treatments are required, but can prove inadequate. Low cardiac output syndrome can quadruple the overall mortality rate for aortocoronary bypass surgery from 2% to 8%. Therefore, an urgent need exists for effective forms of preemptive cardioprotection and antioxidant protection may play a crucial role. Our research into the therapeutic potential of propofol, an intravenous anesthetic with antioxidant properties, could have significant impact on outcome in this select population. The proposed study represents a novel therapeutic approach for the prevention of myocardial ischemia-reperfusion injury in diabetic patients undergoing cardiac surgery with cardiopulmonary bypass.

RESEARCH PLAN

Two blinded, randomized controlled phase II studies will be conducted in patients undergoing primary aortocoronary bypass surgery.

STUDY A

Specific Aims:

1. To determine whether propofol increases nitric oxide bioavailability and decreases ET-1 formation in diabetic patients undergoing aortocoronary bypass surgery
2. To determine whether propofol inhibits superoxide formation or downregulates iNOS gene expression in cardiac tissue.

Hypothesis:

Oxidant stress during myocardial reperfusion promotes the conversion of NO to the cardiotoxic free radical, peroxynitrite, and enhances the formation of the vasoconstrictor ET-1 in diabetic patients. We postulate that these factors cause postoperative cardiac dysfunction of the ischemic-reperfused diabetic heart.

STUDY B

Specific Aim:

To determine whether a high dose of intravenous insulin increases the effect of propofol on perioperative oxidative stress.

Hypothesis: Insulin, by preventing hyperglycemia, enhances propofol's effect on oxidative stress.

Methods

In Study A, 144 patients (72 patients with Type II DM + 72 patients with no DM) will be randomized to receive either propofol 120 ug/kg/min or isoflurane 0.5 to 2% for a treatment interval of 120 to 150 min (10 min before and during CPB, and for 15 min following aortic declamping). All patients will receive a continuous intravenous (I.V.) infusion of insulin as needed to maintain glucose levels at 8 to 12 mmol/L.

In Study B, 72 Type II diabetic patients will be randomized to isoflurane or propofol cardioprotection. All patients will be treated with the perioperative hyperinsulinemic clamp to maintain blood glucose levels within a target range of 4.5 - 6 mmol/L for up to 6 hours following release of aortic crossclamp.

Arterial and coronary sinus blood will be sampled simultaneously before initiation of CPB and at 5 min reperfusion for Troponin I, 15-F2t-isoP, nitrotyrosine and tyrosine, ET-1, and TNF-alpha. An index of myocardial derived 15-F2t-isoP and peroxynitrite will be determined from the Cs-Ao difference in percentage ratio of plasma free 15-F2t-isoP and nitrotyrosine to tyrosine, respectively.

Atrial tissue will be sampled before initiation of CPB and at 15min reperfusion for detection of iNOS, eNOS and superoxide formation. This will coincide with central venous blood sampling for measurement of the concentration of propofol.

The levels of 15-F2t-isoP, nitrotyrosine and tyrosine, ET-1, and TNF-alpha in blood will be determined at 2 hours postoperatively. Troponin I levels will be determined at 2, 12, and 24 hours postoperatively. Cardiac function will be assessed up to 6 hours postoperatively by pulmonary artery catheter and transesophageal echocardiography.

This study represents a novel therapeutic approach for the prevention of myocardial ischemia-reperfusion injury. This study on diabetic patients will provide the prerequisite knowledge for a randomized clinical trial powered to detect clinical outcomes in this high risk patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with and without Type II Diabetes Mellitus
2. Hemodynamically Stable
3. Non urgent Coronary Bypass Grafting utilizing Cardiopulmonary Bypass

Exclusion Criteria:

1. Age less than 18 or greater than 80 years of age
2. refuse informed consent
3. Co-existing valvular heart disease
4. Acute or evolving myocardial infarction
5. hypersensitivity to propofol or formulation component
6. Use of NSAIDs, Vitamins C or E within 5 to 7 days of surgery

Ages: 19 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 137 (Actual)
Dates: Start 2005-04; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Perioperative Plasma 15 f2t isoprostane, a biologically active marker of oxidative stress | 24 hours post operation

SECONDARY OUTCOMES:
Perioperative (includes coronary sinus levels) plasma antioxidant concentration; ET-1, TNF alpha, Troponin I, peroxynitrite; gene and protein expression of eNOS and iNOS; hemodynamics | 24 hours post operation

CONTACTS AND LOCATIONS:
Overall Officials: David M. Ansley, MD, Principal Investigator — University of British Columbia; Peter T. Choi, MD, Study Director — University of British Columbia; David DY Chen, Ph.D, Study Director — University of British Columbia
Locations (1):
- UBC Dept of Anesthesiology, Pharmacology & Therapeutics, Vancouver Acute Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Ansley DM, Raedschelders K, Choi PT, Wang B, Cook RC, Chen DD. Propofol cardioprotection for on-pump aortocoronary bypass surgery in patients with type 2 diabetes mellitus (PRO-TECT II): a phase 2 randomized-controlled trial. Can J Anaesth. 2016 Apr;63(4):442-53. doi: 10.1007/s12630-015-0580-z. Epub 2015 Dec 31. PMID 26721648